CLINICAL TRIAL: NCT04746196
Title: Relationship Between Galectin-3 Level and Disease Activity in Ankylosing Spondylitis Patients
Brief Title: Galectin-3 Level in Ankylosing Spondylitis Patients
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gul Devrimsel, Clinical Professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2016/85
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 45 ankylosing spondylitis patients.: Patients diagnosed with ankylosing spondylitis according to Modified New York criteria were included in the study.
  Interventions: Other: Serum galectin-3 concentration was measured.
- 35 controls: Healthy controls
  Interventions: Other: Serum galectin-3 concentration was measured.

INTERVENTIONS:
Other: Serum galectin-3 concentration was measured. — Serum galectin-3 concentration was measured using a commercial chemiluminescent microparticle immunoassay.

SUMMARY:
Forty-five AS patients and 35 healthy controls were enrolled in this study. Patients diagnosed with AS according to Modified New York criteria were included in the study. Clinical and laboratory measurements, duration of symptoms, age and body mass index (BMI) of AS patients were performed and compared with age and BMI matched control group.

DETAILED DESCRIPTION:
Detailed histories of all participants were obtained, and systemic and rheumatologic examinations were performed. We excluded all participants who had a history of hyperlipidemia, liver, renal, hematological, familial thyroid, neoplastic, autoimmune infectious diseases and receiving anti-inflammatory drugs.

We measured serum galectin-3 levels using a commercial chemiluminescent microparticle immunoassay. The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) was used to assess disease activity in AS patients.

ELIGIBILITY:
Inclusion Criteria:

* Ankylosing spondylitis patients
* Healthy controls

Exclusion Criteria:

* Hyperlipidemia
* Liver diseases
* Renal diseases
* Hematological diseases
* Familial thyroid diseases
* Neoplastic diseases
* Autoimmune infectious diseases
* Receiving anti-inflammatory drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ankylosing spondylitis patients and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Relationship Between Galectin-3 Level and Disease Activity in Ankylosing Spondylitis Patients | 5 months
  Correlation

IPD SHARING:
Plan to Share IPD: Undecided